CLINICAL TRIAL: NCT00975052
Title: A Randomized, Placebo-Controlled, Double-Blind, Double-Dummy, Four-Period Crossover Study to Assess the Effects of Concomitant Administration of MK0431 and Metformin Alone and in Combination on Post-Meal Incretin Hormone Concentrations in Healthy Adult Subjects
Brief Title: A Study of the Effects of Sitagliptin (MK0431) and Metformin on Incretin Hormone Concentrations (0431-050)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-050; MK0431-050; 2009_661
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- A (Active Comparator): Sitagliptin alone
  Interventions: Drug: sitagliptin phosphate
- B (Active Comparator): Metformin alone
  Interventions: Drug: Comparator: metformin
- C (Experimental): Sitagliptin and metformin concomitantly
  Interventions: Drug: Comparator: sitagliptin and metformin
- D (Placebo Comparator): Placebo
  Interventions: Drug: Comparator: placebo

INTERVENTIONS:
Drug: sitagliptin phosphate — 100 mg sitagliptin daily for two days in one out of four treatment periods
  Arms: A
Drug: Comparator: metformin — 500 mg twice daily on Day 1 and 1000 mg once daily on Day 2 in one of four treatment periods.
  Arms: B
Drug: Comparator: sitagliptin and metformin — 100 mg sitagliptin once daily and 500 mg metformin twice daily on Day 1 and 100 mg sitagliptin once daily and 1000 mg metformin once daily on Day 2 in one of four treatment periods.
  Arms: C
Drug: Comparator: placebo — Placebo only on Days 1 and 2 in one of four treatment periods.
  Arms: D

SUMMARY:
This study will determine the effect of concomitant administration of sitagliptin and metformin on post-meal incretin hormone concentrations in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Subject is in good health
* Subject has been a nonsmoker for at least 6 months
* Subject is willing to avoid strenuous activity from the screening visit until the end of the study
* Subject agrees not to consume grapefruit products during the study and to avoid all fruit juices 24 hours before and after study drug administration

Exclusion Criteria:

* Any history of stroke or neurological disorder
* Subject has a history of cardiovascular, blood, endocrine or liver diseases
* Subject has a history of cancer

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2006-01; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Weighted average active GLP-1 (glucagonlike peptide-1) concentrations | 4 hours after the postdose meal

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Migoya EM, Bergeron R, Miller JL, Snyder RN, Tanen M, Hilliard D, Weiss B, Larson P, Gutierrez M, Jiang G, Liu F, Pryor KA, Yao J, Zhu L, Holst JJ, Deacon C, Herman G, Thornberry N, Amatruda J, Williams-Herman D, Wagner JA, SinhaRoy R. Dipeptidyl peptidase-4 inhibitors administered in combination with metformin result in an additive increase in the plasma concentration of active GLP-1. Clin Pharmacol Ther. 2010 Dec;88(6):801-8. doi: 10.1038/clpt.2010.184. Epub 2010 Nov 3. PMID 21048706